CLINICAL TRIAL: NCT05934786
Title: Rehabilitation of Cognition and Psychosocial Well-being - A Better Life With Epilepsy
Brief Title: Rehabilitation of Cognition and Psychosocial Well-being in Epilepsy
Acronym: ReCaPABLE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vilnius University (Other)
Responsible Party: Principal Investigator, Ruta Mameniskiene, Professor, senior researcher, Vilnius University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: ReCaP-ABLE-1
Record Dates: First submitted 2023-06-15; First posted 2023-07-07 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Epilepsy
Keywords: Epilepsy; neuropsychology; memory; cognitive functions; quality of life; mental health; rehabilitation
MeSH Terms: conditions — Epilepsy; Psychological Well-Being | interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early intervention group (Active Comparator): The intervention is planned to consist of six individual one-hour therapy sessions with certified psychologists followed by two group sessions (a total of two months (8 weeks) per patient).
  Interventions: Behavioral: Cognitive rehabilitation
- late intervention group (Active Comparator): For 8 weeks this group will receive the usual treatment, then, after repeated cognitive evaluation, will receive the same intervention: six individual one-hour therapy sessions with certified psychologists followed by two group sessions (a total of two months per patient).
  Interventions: Behavioral: Cognitive rehabilitation

INTERVENTIONS:
Behavioral: Cognitive rehabilitation — Six individual one-hour therapy sessions with certified psychologists followed by two group sessions (a total of two months per patient). The intervention will consist of all parts of the Strategies-Outsourcing-Social support toolbox (Baxendale, 2020) and include psychoeducation, lifestyle issues, coping strategies and homework.

SUMMARY:
Epilepsy is a complex and chronic neurological disorder whose definition is not limited to seizures and also includes social, psychological, and cognitive consequences associated with this frequent condition. Despite good knowledge of the burden of cognitive deficits and psychosocial difficulties in epilepsy, there have been few attempts to address these issues through rehabilitation programs. The Rehabilitation of Cognition and Psychosocial well-being - A Better Life with Epilepsy (ReCaP-ABLE) study will consist of the creation and implementation of a psychological intervention in a randomized waitlist-controlled trial within a sample of adults with epilepsy. The trial is designed to provide novel evidence regarding 1) the effectiveness of a psychological-cognitive intervention in improving quality of life, objective and subjective cognitive functioning as well as reducing mental health symptomatology, 2) the target epilepsy population for which cognitive and psychosocial rehabilitation is most effective, and 3) the transfer effects of such an intervention. This interdisciplinary trial involving neurology and psychology specialists is set to guide evidence-based treatment for cognitive and psychological comorbidities that are prevalent in epilepsy but receive insufficient attention in clinical settings.

DETAILED DESCRIPTION:
The aim of the current project is to conduct a randomized waitlist-controlled trial of an original CoRE program, assess its overall efficacity and determine factors associated with a better response to this intervention.

Work schedule Objective 1: To prepare for the study before patient enrolment (2023-04-01 to 2023-12-31, 9 months) Task 1.1. Acquisition of ethical approval according to local regulations, preparation of infrastructure (e.g., reservation of dedicated examination rooms), and personnel. The required infrastructure for clinical examination and evaluation (e.g., electroencephalography, examination rooms) will be available within the clinical center of Vilnius University Hospital Santaros Klinikos while the infrastructure for the conduct of the intervention will be available at the Counseling and training center of the Faculty of Philosophy at Vilnius University. Vilnius University will also provide access to the data management software "MIDAS" and the statistical package for data analysis (SPSS).

Task 1.2. Development of experimental testing material and intervention. This subtask will be accomplished through meetings between investigators in clinical neurology and psychology. Experimental testing material will be developed after conducting a literature review and discussing the tests' feasibility (e.g., duration, mode of application, result analysis).

Task 1.3. Preparation of the study protocol for publication (expected acceptance before patient enrolment) Objective 2: To start patient enrolment and baseline evaluation (2024-01-01 to 2024-02-31, 2 months) and proceed with continuous enrolment, evaluation, intervention, and follow-up (2024-03-01 to 2024-11-30, 9 months).

Task 2.1. Patient recruitment and baseline evaluation Patients will be recruited by neurologists and explained the purpose and workflow of the trial.

The sample size was calculated for a between-group interaction of a two-way repeated measures analysis of variance (ANOVA) with f=0.40, α=0.05, β=0.95, two groups (early and late intervention), three measurement points, 0.5 correlation between repeated measures and no adjustment for non-sphericity. The resulting sample size of n=58 (G*Power 3.1.9.7) was increased by 20% to n=70 to account for dropouts and corresponded well to the mean sample size and attrition rates in previous trials (Joplin et al., 2018).

Inclusion criteria:

Active epilepsy (medication for epilepsy and/or had at least one seizure in the past year) Adults (>17 years) Lithuanian speaker No intellectual disability

Exclusion criteria:

Sensory or motor deficit preventing task completion Epilepsy surgery planned during the project Active non-paroxysmal comorbid disorder of the central nervous system (e.g., neurodegeneration, multiple sclerosis) Active psychiatric disorder during the past year Psychoactive substance use (except social alcohol, tobacco, and caffeine use)

Components of the baseline evaluation:

Demographic and socioeconomic characteristics (case report form) Clinical characteristics (e.g., seizure frequency, type and duration of epilepsy, medication use, comorbidities, previous exposure to psychological counseling), case report form.

Epilepsy re-evaluation by the neurologist (including electroencephalography) Questionnaire data (scales used): quality of life (QOLIE-31-P), anxiety (GAD-7), depression (NDDI-E), suicidality (Columbia Suicide Severity Rating Scale), metacognition (MCQ-30), Jacoby's 3-item Stigma Scale, antiseizure drug adverse effects (LAEP), the Short Form (36) Health Survey, subjective evaluation of cognitive functions (ad hoc Likert scales 0 to 10).

Objective neuropsychological assessment, up to one hour per examination (indicated examples may be substituted by equivalent tests):

Reaction speed (e.g., Trail Making Tests A and B) Working memory (e.g., Digit Span Test) Verbal fluency (e.g., categorical, phonemic naming) Short-term and long-term memory: verbal (short story or word list) and visuospatial (complex figure) at three delays (e.g., immediate, 30 min, and 4 weeks) to test for accelerated forgetting.

Experimental memory tasks with high everyday significance (e.g., map learning, appointment memory, close autobiographical memory) Task 2.2. The intervention (2024-03-01 to 2024-11-31 (early intervention group) and 2025-06-01 to 2026-03-31 (late intervention group)) Patient randomization will be done using dedicated software (e.g., https://www.randomizer.org/). The investigators performing questionnaire-based and neuropsychological assessment will be blinded from the status of the patient.

The intervention is planned to consist of six individual one-hour therapy sessions with certified psychologists followed by two group sessions (a total of two months per patient). The intervention will consist of all parts of the Strategies-Outsourcing-Social support toolbox (Baxendale, 2020) and include psychoeducation, lifestyle issues, coping strategies and homework. It will be developed after group meetings and all psychologists will be trained by a leading specialist to ensure standardization.

Task 2.3. End of patient recruitment and intervention, last follow-up investigations (2024-12-01 to 2025-03-31, 4 months) Objective 3: To conduct data analysis and disseminate the results (2025-04-01 to 2026-03-31, 12 months) Task 3.1 Data analysis, drafting, and editing of the final report, publication, and presentation of the study results (2025-04-01 to 2026-03-31, 12 months).

The efficacy of the intervention will be defined as a significant improvement in one of the primary outcomes (quality of life or verbal memory), tested with a repeated measure between factors AN(C)OVA. Dynamic changes of other outcome measures will be tested respectively. The association between demographic and clinical variables with study endpoints will be conducted by means of linear and ordinal regression modeling. Open-access publishing of the study results will be sought.

Intervention is simultaneously done for the late intervention group, which is treated as a waitlist control during data analysis (see Task 2.2).

ELIGIBILITY:
Inclusion Criteria:

* Active epilepsy (medication for epilepsy and/or had at least one seizure in the past year)
* Adults (>17 years)
* Lithuanian speaker
* No intellectual disability

Exclusion Criteria:

* Sensory or motor deficit preventing task completion
* Epilepsy surgery planned during the project
* Active non-paroxysmal comorbid disorder of the central nervous system (e.g.,
* neurodegeneration, multiple sclerosis)
* Active psychiatric disorder during the past year
* Psychoactive substance use (except social alcohol, tobacco and caffeine use)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-10-11 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Quality of life index | Immediately before intervention and after.
  QOLIE-31-P will be used before and after interventions. The efficacy of the intervention will be defined as a change from baseline value immediately before intervention at 8 weeks immediately after intervention
Delayed verbal recall | Immediately before intervention, after 30 minutes and after 4 weeks immediately after intervention
  The short story and word list will be used immediately before the intervention, repeated after 30 minutes and immediately after intervention after 4 weeks. The efficacy of the intervention will be defined as a change from baseline value at 30 minutes and a change from baseline value at 4 weeks
Delayed visual recall | Immediately before intervention, at 30 minutes and immediately after intervention at 4 weeks
  The complex figure test will be used immediately before the intervention, repeated after 30 minutes and immediately after intervention after 4 weeks. The efficacy of the intervention will be defined as a change from baseline value at 30 minutes and a change from baseline value at 4 weeks.

SECONDARY OUTCOMES:
Mood | Immediately before and two times (immediately after the intervention and 8 weeks later).
  The Neurological Disorders Depression Inventory for Epilepsy (NDDI-E) for evaluation of depression will be used. The change from baseline value at 8 and 16 weeks will be assessed
Anxiety | Immediately before and after intervention.
  Generalized anxiety disorder (GAD) inventory for evaluation of anxiety will be used two times - before and after interventions (after 8 and 16 weeks). The change from baseline value at 8 and 16 weeks will be assessed
Stigma | Immediately before and after intervention.
  Jacoby's 3-item Stigma Scale will be used two times - before and after interventions (after 8 and 16 weeks). The change from baseline value at 8 and 16 weeks will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Vilnius University Hospital Santaros Klinikos, Vilnius, Lithuania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Puteikis K, Jakoniene A, Jasionis A, Wolf P, Mameniskiene R. Rehabilitation of cognition and psychosocial well-being - a better life with epilepsy (ReCaP-ABLE): a protocol for a randomized waitlist-controlled trial. Front Neurol. 2023 Oct 27;14:1273550. doi: 10.3389/fneur.2023.1273550. eCollection 2023. PMID 37965169